CLINICAL TRIAL: NCT04735900
Title: Detection of Progressive Disease in Metastatic Colorectal Cancer Patients by NPY Methylation in Liquid Biopsies
Brief Title: lead-in FOLICOLOR Trial: Following Therapy Response Through Liquid Biopsy in Metastatic Colorectal Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20/17/224
Record Dates: First submitted 2020-12-30; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- First-line FOLFOX/FOLFIRI and panitumumab. (Experimental): Chemotherapeutic agents will be given as an intravenous infusion at a dose and interval consistent with standard institutional practice.
  Interventions: Procedure: Liquid biopsy sampling

INTERVENTIONS:
Procedure: Liquid biopsy sampling — Biweekly liquid biopsy sampling to measure circulating tumor DNA (ctDNA) level up to and including 9 months after start first-line therapy.

SUMMARY:
Detection of progressive disease by neuropeptide Y (NPY) methylation in liquid biopsies in patients with RAS and BRAF wild-type, unresectable, metastatic colorectal cancer receiving first-line treatment FOLFOX/FOLFIRI and panitumumab.

DETAILED DESCRIPTION:
Prospective, multicentric interventional study to optimize the cutoff value of NPY methylation in liquid biopsies in metastatic colorectal cancer patients treated with first-line FOLFOX/FOLFIRI and panitumumab.

Inclusion is possible after histologically or cytologically proven colorectal adenocarcinoma with metastatic lesions according to RECIST 1.1 at the start of first-line treatment using FOLFOX/FOLFIRI and panitumumab. Patient must have a proven RAS and BRAF wild-type tumor.

Patients will be followed by study protocol up to and including the first CT scan following the last liquid biopsies taken, or when a follow-up period of 11 months is reached, until death, until metastasectomy, until lost to follow-up or until (consent) withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman ≥ 18 years of age at the time the informed consent is obtained
* Eastern cooperative oncology group (ECOG) performance status of 0 or 1
* Histologically or cytologically confirmed adenocarcinoma of the colon or rectum in subjects with unresectable metastatic (M1) disease
* At least 1 uni-dimensionally measurable lesion of at least 10 mm per RECIST 1.1 guidelines using conventional techniques (CT scan). Lesion must not be chosen from a previously irradiated field, unless there has been documented disease progression in that field after irradiation and prior to inclusion. All sites of disease must be evaluated <28 days prior to the start of first-line therapy
* Wild-type RAS tumor status (of tumor tissue)
* Wild-type BRAF tumor status (of tumor tissue)
* Adequate hematologic, renal, hepatic and coagulation function
* Starting a first-line treatment with a combination of FOLFOX/FOLFIRI and panitumumab

Exclusion Criteria:

* History of prior or concurrent central nervous system metastases
* History of other malignancy, except:

  * Malignancy treated with curative intent and with no known active disease present for ≥ 3 years prior to start therapy and felt to be at low risk for recurrence by the treating physician
  * Adequately treated non-melanomatous skin cancer or lentigo maligna without evidence of disease
  * Adequately treated cervical carcinoma in situ without evidence of disease
  * Prostatic intraepithelial neoplasia without evidence of prostate cancer
* Prior chemotherapy or other systemic anticancer therapy for the treatment of metastatic colorectal carcinoma including but not limited to bevacizumab and anti-Epidermal Growth Factor Receptor (EGFR) therapy (e.g. cetuximab, panitumumab, erlotinib, gefitinib, lapatinib)
* Prior adjuvant chemotherapy (including oxaliplatin therapy) or other adjuvant systemic anticancer therapy including but not limited to bevacizumab and anti-EGFR therapy (e.g. cetuximab, panitumumab, erlotinib, gefitinib, lapatinib) for the treatment of colorectal cancer ≤ 6 months prior to start therapy with the following exceptions:

  * Subjects may have received prior fluoropyrimidine therapy if administered solely for the purpose of radiosensitization for the adjuvant or neoadjuvant treatment of rectal cancer
* Radiotherapy ≤ 14 days prior to start therapy. Subjects must have recovered from all radiotherapy-related toxicities.
* Significant cardiovascular risk
* History of interstitial lung disease (e.g., pneumonitis or pulmonary fibrosis) or evidence of interstitial lung disease on diagnostic CT scan
* Active inflammatory bowel disease or other bowel disease causing chronic diarrhea (defined as ≥ Common Terminology Criteria (CTC) grade 2, [Common Terminology Criteria for Adverse Events (CTCAE) version 5.0])
* Peripheral sensory neuropathy (≥ CTC grade 2 [CTCAE version 5.0])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Optimize cutoff value | Start cycle 1 of first-line FOLFOX/FOLFIRI and panitumumab therapy until the day on which the first CT scan is performed following the liquid biopsies taken 9 months after the start of first-line therapy, or when 11 months of follow-up is reached.
  Optimization of the cutoff value for NPY methylation in liquid biopsies (ctDNA) in metastatic colorectal cancer patients receiving first-line FOLFOX/FOLFIRI and panitumumab to discriminate between progressive and non-progressive disease as determined by CT scans based on RECIST criteria 1.1. To this end, a Receiver Operating Characteristic (ROC) curve will be developed with data of this study.

SECONDARY OUTCOMES:
Determine progression free and 9-month survival | Start cycle 1 of first-line FOLFOX/FOLFIRI and panitumumab therapy until the day on which the first CT scan is performed following the liquid biopsies taken 9 months after the start of first-line therapy, or when 11 months of follow-up is reached.
  To determine the progression free and 9-month survival of RAS and BRAF wild-type metastatic colorectal cancer patients. The progression free survival is defined as time from inclusion to the date of first disease progression per RECIST 1.1 criteria, or death. The 9-month survival will be determined as percentage surviving at 9 months after the start of first-line therapy.

OTHER OUTCOMES:
Exploratory objective 1 | Start cycle 1 of first-line FOLFOX/FOLFIRI and panitumumab therapy until the day on which the first CT scan is performed following the liquid biopsies taken 9 months after the start of first-line therapy, or when 11 months of follow-up is reached.
  To compare the use of NPY methylated ctDNA and carcinoembryonic antigen (CEA) to predict progressive disease.
Exploratory objective 2 | Start cycle 1 of first-line FOLFOX/FOLFIRI and panitumumab therapy until the day on which the first CT scan is performed following the liquid biopsies taken 9 months after the start of first-line therapy, or when 11 months of follow-up is reached.
  Further exploration of ctDNA in liquid biopsies and searching for novel biomarkers.
Exploratory objective 3 | Start cycle 1 of first-line FOLFOX/FOLFIRI and panitumumab therapy until the day on which the first CT scan is performed following the liquid biopsies taken 9 months after the start of first-line therapy, or when 11 months of follow-up is reached.
  To assess the quality of life and the patient experience in the patient population with regard to the use of liquid biopsies for follow-up through questionnaires. This will include, but will not be limited to the following: burden of extra blood samples (extra blood samples during routine blood test), burden of CT scan with intravenous contrast, confidence in liquid biopsy guided therapy (ctDNA analysis) compared to CT scan guided therapy and preference between extra blood sample and CT scan (taking into account: burden, pain, time in the hospital, extra travel time to the hospital, confidence in technique…).

CONTACTS AND LOCATIONS:
Overall Officials: Marc Peeters, MD, PhD, Principal Investigator — Antwerp University Hospital (UZA)
Locations (6):
- Belgium (6):
  - AZ Klina, Brasschaat
  - Antwerp University Hospital (UZA), Edegem
  - AZ Maria Middelares, Ghent
  - AZ Groeninge, Kortrijk
  - AZ Nikolaas, Sint-Niklaas
  - GZA, Wilrijk

DOCUMENTS (1):
  • Study Protocol (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT04735900/Prot_000.pdf